CLINICAL TRIAL: NCT02716766
Title: Randomised Phase II Trial of Sorafenib, Capecitabine and Oxaliplatin (SECOX) Versus Single Agent Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Study of SECOX Versus Sorafenib as First-Line Treatment in Patients With Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKU-MONC-HCC-001
Record Dates: First submitted 2016-03-09; First posted 2016-03-23 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Carcinoma, Hepatocellular; Secondary
Keywords: Sorafenib; Drug Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis | interventions — Sorafenib; Capecitabine; Oxaliplatin

ARMS (2):
- SECOX (Experimental): Sorafenib 400 mg twice daily from Day 1 to 14, Capecitabine 850 mg/m2 twice daily from Day 1 to 7, Oxaliplatin 85 mg/m2 on Day 1
  Interventions: Drug: Sorafenib; Drug: Capecitabine; Drug: Oxaliplatin
- Sorafenib (Active Comparator): Sorafenib 400 mg twice daily from Day 1 to 14
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — PO
  Other Names: Nexavar
Drug: Capecitabine — PO
  Other Names: Xeloda
  Arms: SECOX
Drug: Oxaliplatin — IV
  Arms: SECOX

SUMMARY:
The purpose of this study is to determine if sorafenib, capecitabine and oxaliplatin (SECOX) regimen is more effective than sorafenib alone in the treatment of advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic hepatocellular carcinoma (HCC) not suitable for surgery or various loco-regional therapies.
* Diagnosis of HCC confirmed either by cyto-histological confirmation or by non-invasive criteria according to the European Association for Study of Liver disease (EASL) criteria.
* Child-Pugh A or B7 cirrhosis.
* Eastern Co-Operative Group (ECOG) performance status ≤ 2.
* Life expectancy of ≥ 12 weeks.
* Adequate organ function (blood transfusion or use of biologic response modifiers is not permitted).
* Measurable disease with at least one lesion, which is at least 1 cm in one dimension on computed tomography (CT) or magnetic resonance imaging (MRI).
* Able and willing to meet all protocol-required treatments, investigations and visits.
* Signed written informed consent form.

Exclusion Criteria:

* Prior systemic therapy for advanced HCC.
* Central nervous system (CNS) metastasis.
* History of liver transplantation.
* Peripheral sensory neuropathy with functional impairment before the first cycle of treatment.
* History of cardiac disease.
* Uncontrolled hypertension.
* Women who are pregnant or breast-feeding, or women of child-bearing potential who are unable or unwilling to practice a highly effective means of contraception.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | Approximately 18 months
  Time from study treatment to radiological progression

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 18 months
  Proportion of patients with a complete response (CR) or partial response (PR)
Progression-free survival (PFS) | Approximately 18 months
  Time from study treatment to radiological disease progression or death due to any causes
Overall survival (OS) | Approximately 33 months
  Time from study treatment to the date of death due to any cause or last follow-up date
Frequency and severity of adverse events and laboratory abnormalities | Approximately 18 months
  Type, frequency, severity of adverse events (AEs) and laboratory abnormalities as graded by NCI CTCAE v4.03, and their seriousness and relationship to study medications

OTHER OUTCOMES:
Quality of life (QoL) | Baseline, up to approximately 18 months
  Changes in patient-reported QoL status is assessed using EORTC core quality of life questionnaire QLQ-C30 with the HCC-specific module EORTC QLQ-HCC18. EORTC QLQ-HCC18 is an 18-item questionnaire designed to be used along with the 30-item EORTC QLQ-C30. EORTC QLQ-HCC18 questionnaire includes 8 symptom scales such as fatigue, jaundice, nutrition, pain, fever, abdominal swelling, sexual interest, and body image. These scores range from 0-100 for the role functioning scale, physical function scale and the other QLQ-C30 scales and HCC18 symptom complexes.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yau, MD, Study Chair — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No